CLINICAL TRIAL: NCT02782728
Title: Trauma-informed Personalized Scripts (TIPS) to Address Relationship Abuse and Reproductive Coercion in Family Planning Clinics
Brief Title: Trauma-informed Personalized Scripts (TIPS) for Relationship Abuse
Acronym: TIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Elizabeth Miller, Chief of Adolescent Medicine, Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO15080163-02
Record Dates: First submitted 2016-05-12; First posted 2016-05-25 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Violence; Abuse
Keywords: intimate partner violence; reproductive coercion; women's health; relationship abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIPS-Basic (Active Comparator): Providers receive tailored scripts based on the patient's responses to the questions administered via tablet.
  Interventions: Behavioral: TIPS-Basic
- TIPS-Plus (Experimental): Patients receive tailored messages in addition to the scripts given to providers.
  Interventions: Behavioral: TIPS-Plus

INTERVENTIONS:
Behavioral: TIPS-Plus — Patients receive brief psycho-educational messages on a tablet computer following completion of questionnaire about personal experiences of intimate partner violence (IPV), sexual assault (SA), and reproductive coercion (RC). These messages are tailored to each patient and are based on their responses to specific items. The messages serve as prompts to encourage the patient to continue the discussion about various topics (healthy relationships, birth control methods, harm reduction) with their provider during their clinic visit. Simultaneously, providers receive a print out with a series of scripts tailored to the patient's responses to introduce healthy relationships education, brief counseling, and harm reduction.
  Arms: TIPS-Plus
Behavioral: TIPS-Basic — Patients complete tablet questionnaire about personal experiences of IPV/SA/RC and based on responses, providers receive a print out with a series of scripts tailored to the patient's responses to introduce healthy relationships education, brief counseling, and harm reduction.
  Arms: TIPS-Basic

SUMMARY:
This pilot study will evaluate a computer-based intervention titled "Trauma-informed Personalized Scripts" (TIPS). The goal of this intervention is to improve patient-provider communication about sensitive topics such as intimate partner violence (IPV) and reproductive coercion (RC). The main aim of this study is to pilot test TIPS in family planning clinics using a randomized study design to compare the basic version of TIPS (a computer-based assessment with provider scripts only) to an enhanced TIPS containing a tailored brief intervention for patients along with provider scripts. The investigators plan to recruit 240 female patients ages 16-29 for this study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* age 16-29
* English speaking
* Plans to stay in the area for next 6 months

Exclusion Criteria:

* Female clients not of the specified age range.
* Clients who are intoxicated or otherwise not able to provide their own consent will not be eligible to participate.
* Clients who are not able to read English will also be excluded from this pilot study as the survey questions presented via the tablet computer have not been validated yet in any other language.

Ages: 16 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Quality of intervention delivery by provider | Immediately following clinic visit
  Assessment of delivery of brief intervention previously tested and found to be helpful in family planning clinic settings (Addressing Reproductive Coercion in Health Settings (ARCHES), NCT01459458). Summary score based on patient responses on an after-visit exit survey inquiring about what elements of the intervention the provider discussed during clinic visit

SECONDARY OUTCOMES:
Difference in pregnancy risk | baseline to 4 months
  2.1 Change in condom use frequency: Assessment of pregnancy risk reduction through change in frequency of self-reported condom use from baseline to follow-up 2.2 Contraceptive use: Assessment of pregnancy risk reduction through differences in contraceptive use from baseline to follow-up
Change in self-efficacy to enact harm reduction behaviors (mean score) | Baseline to 4 months
  Baseline-adjusted differences in mean post-intervention levels of self-efficacy regarding uptake of harm reduction strategies up to 4 months after baseline clinical encounter
Enacting harm reduction behaviors (summary score) | 4 months
  Summary score of use of any harm reduction strategies, measured by investigator developed items that include a range of harm reduction strategies that women may employ to increase their safety
Change in knowledge of sexual and partner violence related services from baseline to follow up | Baseline to 4 months
  Knowing about specified IPV/SV related services comparing baseline and follow up summary scores
Any use of sexual and partner violence related services | 4 months
  Any use of sexual violence related services (summary score) at 4 month follow up
Change in violence victimization from baseline to follow up | Baseline to 4 months
  Among those reporting exposure to violence (IPV/SV/RC) at baseline, summary score of any recent (past 3 months) violence victimization (including IPV/SV/RC), comparing before intervention to after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Miller E, Decker MR, McCauley HL, Tancredi DJ, Levenson RR, Waldman J, Schoenwald P, Silverman JG. A family planning clinic partner violence intervention to reduce risk associated with reproductive coercion. Contraception. 2011 Mar;83(3):274-80. doi: 10.1016/j.contraception.2010.07.013. PMID 21310291
- [Background] Miller E, Decker MR, McCauley HL, Tancredi DJ, Levenson RR, Waldman J, Schoenwald P, Silverman JG. Pregnancy coercion, intimate partner violence and unintended pregnancy. Contraception. 2010 Apr;81(4):316-22. doi: 10.1016/j.contraception.2009.12.004. Epub 2010 Jan 27. PMID 20227548
- [Background] Miller E, McCauley HL, Tancredi DJ, Decker MR, Anderson H, Silverman JG. Recent reproductive coercion and unintended pregnancy among female family planning clients. Contraception. 2014 Feb;89(2):122-8. doi: 10.1016/j.contraception.2013.10.011. Epub 2013 Dec 10. PMID 24331859
- [Background] Miller E, Tancredi DJ, Decker MR, McCauley HL, Jones KA, Anderson H, James L, Silverman JG. A family planning clinic-based intervention to address reproductive coercion: a cluster randomized controlled trial. Contraception. 2016 Jul;94(1):58-67. doi: 10.1016/j.contraception.2016.02.009. Epub 2016 Feb 15. PMID 26892333
- [Derived] Hill AL, Zachor H, Miller E, Talis J, Zelazny S, Jones KA. Trauma-Informed Personalized Scripts to Address Partner Violence and Reproductive Coercion: Follow-Up Findings from an Implementation Randomized Controlled Trial Study. J Womens Health (Larchmt). 2021 Apr;30(4):604-614. doi: 10.1089/jwh.2020.8527. Epub 2020 Nov 18. PMID 33211607
- [Derived] Hill AL, Zachor H, Jones KA, Talis J, Zelazny S, Miller E. Trauma-Informed Personalized Scripts to Address Partner Violence and Reproductive Coercion: Preliminary Findings from an Implementation Randomized Controlled Trial. J Womens Health (Larchmt). 2019 Jun;28(6):863-873. doi: 10.1089/jwh.2018.7318. Epub 2019 Apr 10. PMID 30969147